CLINICAL TRIAL: NCT06520072
Title: Mobile Apps for Preschool Parents (MAPP) Study
Acronym: MAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Hull (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Pamela Hull, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 93603; 2017-68001-34846 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Obesity, Childhood; Nutrition, Healthy; Physical Inactivity; Sleep, Inadequate
Keywords: Mobile Application; Preschool children; Parents; Parenting; Reading
MeSH Terms: conditions — Pediatric Obesity; Sedentary Behavior; Sleep Deprivation | interventions — Mastication

STUDY DESIGN:
Intervention Model Description: 1. The ORGANIZATION SAMPLE has a 2-arm parallel cluster-randomized control trial design, with an attention control design. The clusters are the partner community-based organizations where participants are recruited/enrolled by study staff. The cluster is the level of randomization (not individuals).
  2. The INDIVIDUAL SAMPLE has a 2-arm parallel randomized control trial design, with an attention control design. The individual parent/guardian as the level of randomization (no clusters). After completing the Baseline Survey (Parts 1 and 2), each individual parent/guardian will be randomized to the Intervention Arm or Control Arm.
  Both: Parents/guardians will be asked to use the assigned app for 8-weeks. Next, they will complete the Follow Up Survey, then they have the option to download the other app, if interested. For both arms, usage of the CHEW app will be tracked for up to 20 weeks after the date of study enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm: Nutrition and wellness app (Experimental): The parents/guardians in this study arm will use the Children Eating Well (CHEW) mobile app focused on child and family nutrition and wellness for the first 8 weeks of the study. This app is designed to help parents/guardians of preschool-aged children to improve nutrition, physical activity, sleep, feeding children at mealtimes, and related wellness topics.
  Interventions: Behavioral: Children Eating Well (CHEW) mobile app
- Attention Control Arm: Reading app (Active Comparator): The parents/guardians this study arm will use the Beanstack mobile app (or the Bookroo app, as an alternative) focused on parents reading to their children for the first 8 weeks of the study. This app may help parents/guardians to read more to their preschool children (and other children), which is good for child learning and development.
  Interventions: Behavioral: Beanstalk mobile app

INTERVENTIONS:
Behavioral: Children Eating Well (CHEW) mobile app — The target users of the CHEW app are parents/guardians of preschool aged children. The purpose of the CHEW app is to provide parents/guardians with easy, practical ways to improve nutrition and wellness among their preschool-aged children. The app provides guided goal setting and tracking tools. Parents/guardians set goals related to their preschool-aged children focused on nutrition, physical activity, sleep behaviors and parenting styles. The parents/guardians can also to set goals for themselves for behaviors related to nutrition, physical activity, sleep, and stress. The app does not have features that target children as users.
  The CHEW app was developed by the study team and can be downloaded for mobile devices (phones or tablets) at no cost in the Apple App Store (iOS/Apple) and the Google Play Store (Android). After downloading the CHEW app, enrolled participants must enter the Access Code provided by the study team in order to unlock the app and use it.
  Arms: Intervention Arm: Nutrition and wellness app
Behavioral: Beanstalk mobile app — Beanstack is free commercially-available mobile app that provides goal setting and tracking tools similar to the CHEW app, but focused on a different topic, specifically encouraging parents/guardians to read to their preschool children more frequently. In the case that a parent/guardian is not able to successfully download Beanstack to their mobile device, as a backup alternative they will be asked to use a similar free commercially-available mobile application called Bookroo.
  Beanstack is available to the public for mobile devices (phones or tablets) at no cost in the Apple App Store (iOS/Apple) and the Google Play Store (Android). Bookroo is a web-based application that users access via the mobile device's web browser and looks and functions like a regular mobile application. It should work on any mobile device with a browser and data/wifi access,
  Other Names: Alternative: Bookroo mobile app
  Arms: Attention Control Arm: Reading app

SUMMARY:
The purpose of Mobile Apps for Preschool Parents (MAPP) Study is to test the effectiveness of two mobile applications for parents of preschool aged children: 1) an app focused on child and family nutrition and wellness, and 2) an app focused on parents reading to their children.

DETAILED DESCRIPTION:
The Mobile Apps for Preschool Parents (MAPP) Study addresses an important gap in the scientific literature, which is the need to evaluate the use of parent-targeted, guided goal-setting for childhood obesity risk reduction via a mobile application, specifically for parents of preschool-aged children for early intervention.

Obesity is a leading cause of multiple chronic diseases, including 13 types of cancer, heart disease, stroke, and type II diabetes. Major behavioral determinants of obesity are also independent risk factors for these chronic diseases, including unhealthy diet, lack of physical activity, and poor sleep quality. Childhood obesity increases risk for adult obesity and early onset of conditions such as high blood pressure, high cholesterol, asthma, sleep apnea, and joint problems. Childhood obesity disproportionately affects children of lower socioeconomic status, racial/ethnic minority groups, and rural areas, thus exacerbating and contributing to health disparities among obesity-related health conditions. Children in low-income families that qualify for income-based public assistance programs represent a population that is at high risk for obesity. These programs include the Women, Infants and Children (WIC) Supplemental Nutrition Program; Head Start (preschool child care centers); the Supplemental Nutrition Assistance Program (SNAP); Temporary Assistance for Needy Families (TANF); and Medicaid.

With the Attention Control Arm, the MAPP Study will also contribute valuable information about the effectiveness of using a mobile application with parent-targeted, guided goal-setting for reading to preschool-aged children. Previous studies have shown that adults reading to children is beneficial for child learning and development.

All parents/guardians (both samples and both arms) will be asked to use the respective apps for an 8-week intervention period. The primary outcome will be measured in the Baseline Survey and a Follow Up Survey after completing the 8-week intervention period. After completion of the Follow Up Survey, parents/guardians will be given the option to download and use the other app, if they are interested (i.e., information about the CHEW app for the Control Arm, and information about the Control app for the Intervention Arm). For both the Intervention Arm and those who choose to download the CHEW app in the Control Arm, usage of the CHEW app (i.e., app analytics) will be tracked for up to 20 weeks after the date of study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Guardian (age 18+ years) of a 2-5 year old
* Living in United States
* Receives services at partner community organization (Organization Sample only)

Exclusion Criteria:

* Does not own iOS/Apple or Android mobile device (phone or tablet)
* Does not have internet access for the mobile device (data plan on device or in-home WiFi)
* Not able to successfully load and access the Intervention Arm or Attention Control Arm mobile app on the mobile device at the time of enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Healthy Kids childhood obesity risk score | 2 months
  Using the 19-item Healthy Kids scale, each item is coded from 1 to 5, with 1 being the least healthful and 5 being the most healthful. To calculate the childhood obesity risk score, all 19 items are summed together, ranging from 19 to 95, with higher values reflecting a more healthful, or positive, outcome.

SECONDARY OUTCOMES:
Child intake of sugar-sweetened beverages (Healthy Kids items) | 2 months
  Child intake of sugar-sweetened beverages (Healthy Kids items)
Child intake of fruits and vegetables (Healthy Kids items) | 2 months
  Child intake of fruits and vegetables (Healthy Kids items)
Child intake of energy dense food/beverages (Healthy Kids items) | 2 months
  Child intake of energy dense food/beverages (Healthy Kids items)
Child intake of dairy/calcium (Healthy Kids items) | 2 months
  Child intake of dairy/calcium (Healthy Kids items)
Child physical activity and sedentary behavior (Healthy Kids items) | 2 months
  Child physical activity and sedentary behavior (Healthy Kids items)
Sleep: Child bedtime (Healthy Kids item) | 2 months
  Child bedtime (Healthy Kids item)
Family meals: Eating meals with child (Healthy Kids item) | 2 months
  Eating meals with child (Healthy Kids item)
Child dietary intake (Healthy Kids items) | 2 months
  Child dietary intake (Healthy Kids items)
Diet quality: Variety of child vegetable intake (My Veggies questionnaire) | 2 months
  Variety of child vegetable intake (My Veggies questionnaire)
My Child at Mealtime questionnaire | 2 months
  My Child at Mealtime questionnaire measures food-related parenting styles.
Home Inventory Describing Eating and Activity (Home-IDEA2, food section) | 2 months
  Home Inventory Describing Eating and Activity (Home-IDEA2, food section) measures home food environment.
Frequency of reading to child | 2 months
  Frequency of reading to child
Length of time reading to child | 2 months
  Length of time reading to child

CONTACTS AND LOCATIONS:
Overall Officials: Pamela C Hull, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States